CLINICAL TRIAL: NCT05026944
Title: Effects of Percussive Massage Treatment With Theragun on Pain and Muscle Length on Post Exercise Delayed Onset Muscle Soreness of Calf Muscles
Brief Title: Effects of Percussive Massage Treatment With Theragun on Post Exercise Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/0410 Mahnoor
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Theragun; Percussion; Stretching Exercise; Muscle soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Percussive massage and static stretching exercises
  Interventions: Other: Percussive massage and static stretching exercises
- Group B (Other): Static stretching exercises
  Interventions: Other: static stretching exercises

INTERVENTIONS:
Other: Percussive massage and static stretching exercises — All the study participants will perform 15 minutes treadmill, 15 minutes stationary bicycle at day one. After 24 hours participants with positive DOMS will be treated with 5 minutes of percussive massage and 5 minutes of static stretching exercises. The group will be assessed on Numeric Pain Rating Scale and Short-Form McGill Pain Questionnaire for pain and degree of passive ankle dorsi flexion for calf muscle length at baseline before intervention and immediate 24 hours, 48 hours and 72 hours after the completion of treatment session.
  Arms: Group A
Other: static stretching exercises — All the study participants will perform 15 minutes treadmill, 15 minutes stationary bicycle at day one. After 24 hours participants with positive DOMS will be managed with 5 minutes of static stretching exercises only. The group will be assessed on Numeric Pain Rating Scale and Short-Form McGill Pain Questionnaire for pain and degree of passive ankle dorsi flexion for calf muscle length at baseline before intervention and immediate 24 hours, 48 hours and 72 hours after the completion of treatment session.
  Arms: Group B

SUMMARY:
This project will be Randomized control trial conducted to check the effects of percussive massage treatment with theragun on pain and muscle length on post exercise delayed onset muscle soreness (DOMS) of calf muscles in healthy population so that we can have best treatment option for people with delayed onset muscle soreness, duration will be of 6months,purposive sampling will be done, subject following eligibility criteria from kasrat health and fitness club, will randomly allocated in two groups, baseline assessment will be done, group A will be treated with 5 minutes of percussive massage and 5 minuties of static stretching exercises, while group B will be managed with 5 minutes of static stretching exercises only. Assessment will be done via, Numeric Pain Rating Scale(NPRS), Short-Form McGill Pain Questionnaire (SF-MPQ) and goniometric measurements of passive ankle dorsi flexion for calf muscle length at baseline before intervention and immediately post intervention data will be analyzed by using SPSS version 25

DETAILED DESCRIPTION:
Percussive therapy is a form of soft tissue manipulation the same thing that a massage therapist does during a massage, and is intended to reduce muscle soreness and increase muscle length. The aim of the current study is to determine the effects of percussive massage with theragun and static stretching exercises on muscle length and pain of calf muscles on post exercise (DOMS) delayed onset muscle soreness. It will be a randomized control trail, where initial screening will be done as per the inclusion criteria of healthy female gym users with minimum one week of joining time and developed post-exercise DOMS and ages ranged from 20 to 30 years. Participants with the history of lower leg injuries, any type of neuromuscular disorder and elite level of fitness will be excluded. All the study participants will perform 15 minutes treadmill, 15 minutes stationary bicycle at day one. After 24 hours participants with positive DOMS will be randomly place into experimental and control groups. Experimental group will be treated with 5 minutes of percussive massage and 5 minutes of static stretching exercises, while the control group will be managed with 5 minutes of static stretching exercises only. Participants in both the groups will be assessed on Numeric Pain Rating Scale and Short-Form McGill Pain Questionnaire for pain and degree of passive ankle dorsi flexion for calf muscle length at baseline before intervention and immediate 24 hours, 48 hours and 72 hours after the completion of treatment session.

ELIGIBILITY:
Inclusion Criteria:

Healthy Females will be included Participant's age will be between of 20-30 years Who develops post exercise DOMS after 15 minutes treadmill, 15 minutes stationary bicycle

Exclusion Criteria:

Subject with history of lower extremity injuries Any history type of muscular disorder Elite level of fitness excluded in this study

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd day
  Changes from base Line Numeric Pain Rating Scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain.
SF-MPQ | 3rd day
  The SF-MPQ is a self- reported measure of pain. It assesses both the quality and intensity of subjective pain. The short- form McGill Pain Questionnaire consists of 15 descriptors of pain including 11 from sensory categories and 4 from affective categories.
Goniometer | 3rd day
  A goniometer is an instrument which measures the available range of motion at a joint.
  (To measure ankle dorsi flexion for calf muscle length.)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- KASRAT (Health & Fitness Club), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen LL, Jay K, Andersen CH, Jakobsen MD, Sundstrup E, Topp R, Behm DG. Acute effects of massage or active exercise in relieving muscle soreness: randomized controlled trial. J Strength Cond Res. 2013 Dec;27(12):3352-9. doi: 10.1519/JSC.0b013e3182908610. PMID 23524365
- [Background] Xie Y, Feng B, Chen K, Andersen LL, Page P, Wang Y. The Efficacy of Dynamic Contract-Relax Stretching on Delayed-Onset Muscle Soreness Among Healthy Individuals: A Randomized Clinical Trial. Clin J Sport Med. 2018 Jan;28(1):28-36. doi: 10.1097/JSM.0000000000000442. PMID 28742609
- [Background] Lewis PB, Ruby D, Bush-Joseph CA. Muscle soreness and delayed-onset muscle soreness. Clin Sports Med. 2012 Apr;31(2):255-62. doi: 10.1016/j.csm.2011.09.009. Epub 2011 Nov 23. PMID 22341015
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Ekstrand J, Hagglund M, Walden M. Epidemiology of muscle injuries in professional football (soccer). Am J Sports Med. 2011 Jun;39(6):1226-32. doi: 10.1177/0363546510395879. Epub 2011 Feb 18. PMID 21335353
- [Background] Imtiyaz S, Veqar Z, Shareef MY. To Compare the Effect of Vibration Therapy and Massage in Prevention of Delayed Onset Muscle Soreness (DOMS). J Clin Diagn Res. 2014 Jan;8(1):133-6. doi: 10.7860/JCDR/2014/7294.3971. Epub 2014 Jan 12. PMID 24596744
- [Background] Han JH, Kim MJ, Yang HJ, Lee YJ, Sung YH. Effects of therapeutic massage on gait and pain after delayed onset muscle soreness. J Exerc Rehabil. 2014 Apr 30;10(2):136-40. doi: 10.12965/jer.140106. eCollection 2014 Apr. PMID 24877051
- [Background] Garcia-Sillero M, Benitez-Porres J, Garcia-Romero J, Bonilla DA, Petro JL, Vargas-Molina S. Comparison of Interventional Strategies to Improve Recovery after Eccentric Exercise-Induced Muscle Fatigue. Int J Environ Res Public Health. 2021 Jan 14;18(2):647. doi: 10.3390/ijerph18020647. PMID 33466606
- [Background] Hernandez FA. Effects of Percussion Therapy (Theragun™) on Range of Motion and Athletic Performance: California State University, Long Beach; 2020.
- [Background] Konrad A, Glashuttner C, Reiner MM, Bernsteiner D, Tilp M. The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance. J Sports Sci Med. 2020 Nov 19;19(4):690-694. eCollection 2020 Dec. PMID 33239942
- [Background] Kujala R, Davis C, Young L, editors. The effect of handheld percussion treatment on vertical jump height. International Journal of Exercise Science: Conference Proceedings; 2019.